CLINICAL TRIAL: NCT06832566
Title: Ramadan Fasting Outcomes in Patients With Secondary Adrenal Insufficiency Before and After the Treatment of Hypotension.
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hopital La Rabta (Other)
Responsible Party: Principal Investigator, Melika Chihaoui, Professor, Hopital La Rabta
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LaRabtaEndocrine1/2025
Record Dates: First submitted 2025-02-07; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Secondary Adrenal Insufficiency; Hypotension
Keywords: secondary adrenal insufficiency; intermittent fasting; complications; hypotension; fludrocortisone; quality of life
MeSH Terms: conditions — Hypotension; Intermittent Fasting

STUDY DESIGN:
Intervention Model Description: Prospective, interventional, before/after study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with secondary adrenal insufficiency and hypotension treated with fludrocortisone 0.05mg/d (Experimental): Patients with secondary adrenal insufficiency and hypotension treated with fludrocortisone 0.05mg/day during Ramadan fasting 2025.
  Interventions: Drug: Fludrocortisone 0.1 Milligrams (mg)

INTERVENTIONS:
Drug: Fludrocortisone 0.1 Milligrams (mg) — Treatment of hypotension with fludrocortisone 0.05mg/day in patients with secondary adrenal insufficiency before Ramadan fasting. Outcomes (number of fasted days and complications during fasting) will be compared between Ramadan fasting 2025 (with fludrocortisone) and Ramadan 2023 (without fludrocortisone).

SUMMARY:
Intermittent fasting in patients with adrenal insufficiency is associated with an increased risk of complications, such as dehydration. A recent study showed that nearly half the patients had hypotension before the fasting month and half had signs of dehydration during fasting. So, we are planning to carry out this prospective interventional study in patients with SAI and hypotension to evaluate the effect of treating hypotension with fludrocortisone on the risk of complications during fasting. Patients with secondary adrenal insufficiency and hypotension and who are willing to fast during Ramadan 2025 will be included. Before Ramadan, they will be treated with fludrocortisone at a dose of 50micg/day. The occurrence of complications and the number of fasted days during Ramadan 2025 will be reported and compared with those of Ramadan 2023.

DETAILED DESCRIPTION:
Intermittent fasting during Ramadan is practised by more than one billion people worldwide. Patients with adrenal insufficiency are at risk of complications during fasting. The most frequently reported complications were intense asthenia (88.5%), signs suggestive of dehydration (49.2%), intense thirst (32.8%), and signs of hypoglycaemia (18%) Chihaoui M, et al, Endocrine 2017;55:289-295. https://doi.org/10.1007/s12020-016-1186-0). A recent study showed that lifestyle measures and drug adjustment enabled more patients to fast and reduced the frequency of complications. It also showed that nearly half the patients had hypotension before the fasting month and half had signs of dehydration during fasting (ClinicalTrials.gov ID: NCT05827965 ; Chihaoui et al, Nutrition, 2025; https://doi.org/10.1016/j.nut.2025.112688).

The objective of the study is to compare the number of fasted days and the prevalence of complications during Ramadan fasting in patients with SAI before (2023) and after the treatment of hypotension with fludrocortisone (2025).

Keywords: secondary adrenal insufficiency; intermittent fasting; complications; hypotension; fludrocortisone; quality of life

Type of study: Prospective, interventional, before/after study

Study population:

The study will include patients with SAI and hypotension who participated in our former study in 2023 (ClinicalTrials.gov ID: NCT05827965 ; Chihaoui et al, Nutrition, 2025; https://doi.org/10.1016/j.nut.2025.112688). Patients will be included before the month of Ramadan, from February 15th to February 25th, 2025, according to the following selection criteria:

Inclusion criteria:

* Patients aged over 18 years
* Secondary adrenal insufficiency patients
* Substituted with glucocorticoids for more than one year.
* Participated in the former study in 2023.
* Willing to fast during the month of Ramadan 2025.

Exclusion criteria: cardiac, respiratory, hepatic or renal insufficiency (creatinine clearance < 60 ml/min/1.73m2), advanced neoplasia, undernutrition, diabetes insipidus, diabetes mellitus, neuro-psychiatric disease, infectious or chronic inflammatory disease, hyperthyroidism, uncontrolled hypothyroidism, alcoholism, diuretic intake, glucocorticoid treatment for purposes other than substitution, enzyme inducers, pregnancy, breastfeeding, consent withdrawn, study discontinuation.

Study period: February 15th -April 15th. Ramadan starts on March 1st and ends on March 29th, 2025.

Methods Before Ramadan 2025, patients meeting the inclusion criteria will be enrolled. All patients have to sign a written informed consent.

During the first visit (two weeks before Ramadan), the following data will be recorded:

* gender, age, medical and surgical history, current treatments, medication schedule,
* Physical examination data: weight, height, lying and standing blood pressure.
* Some data will be taken from the medical file: other affected pituitary axes, etiology of the SAI, baseline cortisol, and plasma creatinine.
* Data about 2023 fast (number of fasted days, complications (type, days, time, breaking of the fast (yes/no) will collected from our former study.

Fludocortisone at a dose of 50 micg/day will be added to the treatment of the patients.

During the second visit (one week before Ramadan), the quality of life questionnaire (AddiQoL) will be administered to the patients, blood pressure will be measured, and a blood sample will be collected for the measurement of sodium, potassium and urea.

Throughout Ramadan 2025, patients will have to fill in forms indicating the fasted days and the occurrence of complications (type, time, and break of the fast). Patients will be asked to respond to the AddiQoL questionnaire again during the third week of Ramadan.

Throughout the study, regular telephone contact with one of the investigators will be maintained for any additional information, advice or therapeutic adjustment.

After Ramadan, filled addiQoL questionnaires and forms will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years
* Secondary adrenal insufficiency patients
* Substituted with glucocorticoids for more than one year.
* Participated in the former study in 2023.
* Willing to fast during the month of Ramadan 2025.

Exclusion Criteria:

* cardiac, respiratory, hepatic or renal insufficiency (creatinine clearance < 60 ml/min/1.73m2), advanced neoplasia, undernutrition, diabetes insipidus, diabetes mellitus, neuro-psychiatric disease, infectious or chronic inflammatory disease, hyperthyroidism, uncontrolled hypothyroidism, alcoholism, diuretic intake, glucocorticoid treatment for purposes other than substitution, enzyme inducers, pregnancy, breastfeeding.
* consent withdrawn, study discontinuation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
number of fasted days | One month
  Total days fasted during the month of Ramadan 2025

SECONDARY OUTCOMES:
complications during fasting | One month
  signs of hypotension, dehydration, hypoglycemia..

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital La Rabta, Tunis, Tunisia, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chihaoui et al, Nutrition, 2025; https://doi.org/10.1016/j.nut.2025.112688